CLINICAL TRIAL: NCT06830252
Title: A Randomised Controlled Trial To Evaluate the Effects of Marked Weight Loss Combined With Exercise Training on Metabolic, Immunological, and Imaging Biomarkers of Systemic and Brain Inflammation in Participants Undergoing Bariatric Surgery
Brief Title: Neurological Impact of Weight Reduction and Fitness Interventions
Acronym: NeuroFit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Washington University School of Medicine (Other); Sydney Local Health District (Other Government); Northern Sydney Local Health District (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: X24-0053; ACTRN12624001065583 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2025-01-30; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Overweight
Keywords: Obesity; Bariatric Surgery; Exercise; Neuroinflammation; Cognitive Function
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Neuroinflammatory Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Control participants will undergo bariatric surgery and receive usual clinical care which includes continued communication and reviews from their health team. Control participants will also be given a Fitbit device and have once a month phone follow-up with the study team and Accredited Exercise Physiologist (AEP). The discussion will be based on current literature on exercise for bariatric surgery patients and will not be personalised.
- Excercise (Experimental): Eligible participants will undergo either gastric bypass or gastric sleeve surgery. Between weeks 6 and 18, participants will attend a supervised physical activity programme. This programme will be individualised per each participant's baseline activity and injuries. Participants will attend 2-3 1-hour appointments per week with their Accredited Exercise Physiologist (AEP), The supervised sessions will be delivered either in an individual setting or in a group of up to three, as needed. Following the supervised period, participants will be given an individualised home based programme and will be monitored via the Fitbit and regular phone follow-up till 12-months post-surgery. If participants are not meeting exercising as per their programme, they will be contacted using the escalating methods of email, text message or phone calls and will be invited to attend in-person supervised sessions.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise.
  Arms: Excercise

SUMMARY:
This study will test how significant weight loss through bariatric surgery, combined with a personalised exercise program, affects brain inflammation. Th investigators want to understand the connection between obesity-related body inflammation, metabolic issues, and brain inflammation and function.

DETAILED DESCRIPTION:
This randomised controlled trial aims to evaluate the effects of marked weight loss, via bariatric surgery, combined with a personalised exercise intervention on markers of brain inflammation. This study will allow the investigators to explore the link between excessive adiposity-induced systemic chronic inflammation, metabolic abnormalities, and neuroinflammation. The investigators hypothesise that bariatric surgery, i.e., marked weight loss, and exercise will result in attenuated neuroinflammation (as measured by neuroimaging), improvements in cognitive function, improvements in immune-inflammatory markers, and improvements in cardiometabolic biomarkers at 12 months compared to control.

This study is a parallel group, randomised controlled trial. A 1:1 allocation ratio will be applied to either the intervention group (bariatric surgery and usual care with exercise) or control group (bariatric surgery and usual care). Participants in both arms will be followed over a period of 12 months after surgery. A comprehensive set of evaluations will be performed prior to the surgery, with follow-up in-person evaluations at 6 weeks and 3, 4.5, 6, and 12 months.

The primary objective is to evaluate the effect of bariatric surgery and exercise on neuroinflammation compared to control at 12-months. This will be assessed via a novel neuroimaging technique. Secondary and exploratory objectives are to evaluate the effect of bariatric surgery and exercise on brain structure, cognition, immune-inflammatory markers, cardiometabolic markers, psychosocial factors, diet, and physical functioning compared to control. The investigators would also like to explore within-group differences for all the above from baseline to 12-months.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age.
* Eligible for bariatric surgery.
* Willingness to provide informed consent and willingness to participate and comply with the study requirements

Exclusion Criteria:

* Unable to undertake MRI due to size restrictions i.e., shoulder width more than 70 cm.
* History or clinical manifestation of any other significant metabolic, hematologic, pulmonary, cardio- vascular, gastrointestinal, neurologic, immune, hepatic, renal, urologic, muscular, and joint disorders, or cancer that, in the opinion of the investigator, would make the candidate ineligible for the study. For example, significant joint pain could interfere with adherence to the exercise program.
* Have objectively assessed cognitive impairment as assessed by the Montreal Cognitive Assessment (MoCA) i.e., total score less than 26.
* Non-MRI-compatible implanted devices or implants.
* Inability to exercise via supine ergometer.
* Claustrophobia.
* Psychiatric or behavioural problems (history of drug and alcohol abuse, eating disorder).
* Breastfeeding or pregnant women, or those intending to become pregnant before the scheduled end of the intervention.
* Unwilling to be assigned at random to the exercise or control intervention.
* Unwilling or unable to adhere to the rigors of the exercise intervention or evaluation schedule over the entire one-year period.
* Concurrent participation in any other interventional study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Markers of neuroinflammation | Baseline and 12 months after surgery.
  Between intervention and control at 12 months after surgery. Assessed via DBSI-MRI.

SECONDARY OUTCOMES:
Cognitive function | Baseline, 6 and 12 months after surgery.
  This will be a composite outcome. Validated questionnaires such as Stroop Test.
Anthropometric measures including height (cm), body mass (kg), body mass index (BMI; kg/m2) | Baseline, 6 weeks, 3, 4.5, 6, and 12 months after surgery.
  This will be assessed as a composite outcome. Assessed via a wall-mounted stadiometer and digital scales.
Metabolic biomarkers (e.g., LDL Cholesterol), peripheral blood cell profiling (e.g., WBC), and immune biomarkers (e.g., IL-6) | Baseline, 6 weeks, 3, 4.5, 6, and 12 months after surgery.
  Venous blood collection, analysed via ELISA.
Brain volumes | Baseline and 12 months after surgery.
  Between groups and within groups at 12 months after randomisation with respect to baseline. Assessed via T1 and T2 MRI.

OTHER OUTCOMES:
Flow-mediated dilatation (FMD; %) | Baseline, 4.5, 6, and 12 months after surgery.
  Assessed via high-resolution ultrasound and semi-automated edge detection software.
Carotid intima-media thickness (cIMT; mm) | Baseline and 12 months after surgery.
  Assessed via high-resolution ultrasound and semi-automated edge detection software.
Pulse wave velocity (PWV; m/s) | Baseline, 6 weeks, 3, 4.5, 6, and 12 months after surgery.
  Assessed via the SphygmoCor XCEL System.
Augmentation Index (AI) | Baseline, 6 weeks, 3, 4.5, 6, and 12 months after surgery.
  Assessed via the SphygmoCor XCEL System.
Peripheral and Central blood pressures (mmHg) | Baseline, 6 weeks, 3, 4.5, 6, and 12 months after surgery.
  Assessed via the SphygmoCor XCEL System.
Heart rate variability (HRV; ms2) | Baseline, 6 weeks, 3, 4.5, 6, and 12 months after surgery.
  This will be assessed as a composite outcome. Assessed via the Human Non-Invasive Blood Pressure System.
Bone mineral density (g/cm2) of the hip | Baseline and 12 months after surgery.
  Assessed via the Hologic Discovery W Dual Energy X-Ray (DEXA) Absorptiometry Scanner.
Whole body fat-free mass (%) | Baseline and 12 months after surgery.
  Assessed via the Hologic Discovery W Dual Energy X-Ray (DEXA) Absorptiometry Scanner.
Total sleep time (mins) | Baseline and 12 months after surgery.
  Assessed via the Nox-T3+ Device.
Sleep efficiency (%) | Baseline and 12 months after surgery.
  Assessed via the Nox-T3+ Device.
Sleep-behaviours | Baseline and 12 months after surgery.
  Assessed via validated questionnaires (STOP BANG, SAGIC, and Epworth Sleepiness Scale).
Composite metabolic control | Baseline.
  Glucose and insulin response to oral glucose tolerance test (75g) at 0, 30, 60, 120 minutes.
Diet quantity and quality | Baseline, 6 and12 months after surgery.
  This will be assessed as a composite outcome. This will be assessed via a 3-day Food Diary, analysed with FoodWorks.
Changes in health-related quality of life | Baseline and 12 months after surgery.
  The Medical Outcomes Study Short-Form 36 Health Status Survey (SF-36). The scores will be standardised according to the normative values for the Australian context.
Changes in social-related quality of life | Baseline and 12 months after surgery.
  The Australian version of the Assessment of Quality of Life (AQoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Perkins Centre Clinic, Royal Prince Alfred Hospital, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data collected for the study, including individual patient data and a data dictionary that defines each field in the data set, will be made available as de-identified participant data to researchers who propose to use the data for individual patient data meta-analysis. Data will be shared following approval of the proposal by the corresponding author and a signed data access agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All IPD data arising from the trial will be shared two years after publication of the main results.

REFERENCES:
- [Background] Samara A, Murphy T, Strain J, Rutlin J, Sun P, Neyman O, Sreevalsan N, Shimony JS, Ances BM, Song SK, Hershey T, Eisenstein SA. Neuroinflammation and White Matter Alterations in Obesity Assessed by Diffusion Basis Spectrum Imaging. Front Hum Neurosci. 2020 Jan 14;13:464. doi: 10.3389/fnhum.2019.00464. eCollection 2019. PMID 31992978